CLINICAL TRIAL: NCT06381921
Title: OIME - Objective Integrated Multimodal Electrophysiological Index for the Quantification of Visceral Pain
Brief Title: Objective Integrated Multimodal Electrophysiological Index for the Quantification of Visceral Pain
Acronym: OIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Hugo Posada-Quintero, Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B2023-0046
Record Dates: First submitted 2024-04-17; First posted 2024-04-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Abdominal Pain
Keywords: visceral pain; irritable bowel syndrome; autonomic and muscular activities; biosignals; personalized pain self-management
MeSH Terms: conditions — Abdominal Pain; Visceral Pain; Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: randomized controlled ambulatory trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IBS-PPSM intervention group (Experimental): After the baseline visit, the IBS-PPSM group will receive 10 video modules focused on IBS knowledge and self-management skills plus one-on-one consultation with a nurse for personalized advice about self-monitoring, diet, sleep, and goal setting. The IBS-PPSM group will be taught to use the abdominal belt/smart watch system for daily recording of bio-signals and voluntary report of episodes of visceral pain. We will follow up with all participants 4 weeks after enrollment, in a final lab visit, and measure primary outcomes to compare to the baseline data.
  Interventions: Behavioral: IBS-PPSM intervention
- IBS-control group (No Intervention): The IBS-control group will not receive pain self-management intervention. Participants will be taught to use the abdominal belt/smart watch system for daily recording of bio-signals and voluntary report of episodes of visceral pain. We will follow up with all participants 4 weeks after enrollment, in a final lab visit, and measure primary outcomes to compare to the baseline data.

INTERVENTIONS:
Behavioral: IBS-PPSM intervention — IBS-PPSM intervention includes 10 video modules focused on IBS knowledge and self-management skills plus one-on-one consultation with a nurse for personalized advice about self-monitoring, diet, sleep, and goal setting.
  Arms: IBS-PPSM intervention group

SUMMARY:
The objectives of the study are to 1) Conduct telemetric biosignals (EDA, ECG, and EMG) recording in healthy controls and IBS participants experiencing cutaneous and visceral pain; and 2) Validate the OIME index as a biomarker for quantifying pain in IBS participants and its capability to assess the treatment of IBS pain via an ambulatory trial.

DETAILED DESCRIPTION:
In part 1, data collection for training the OIME model, we will collect autonomic and muscular activities with integrated biosignal device and visceral pain level in both healthy controls and IBS participants. These data will be used to train a machine learning model to produce an objective integrated multimodal electrophysiological (OIME) index.

In part 2, the ambulatory trial, we will collect data to validate the OIME index as a biomarker of pain in IBS participants. We will run an ambulatory trial to validate the OIME index as a biomarker to assess the treatment of IBS pain.

ELIGIBILITY:
Inclusion Criteria:

* Participants need to be diagnosed with IBS by a healthcare provider according to Rome-III or -IV criteria, with a current report of abdominal pain.
* Men and women 18-50 years old
* Able to read and speak English
* Daily access to a computer with internet access.

Exclusion Criteria:

* Other chronic pains that are usually not comorbid with IBS, e.g., diabetic neuropathy, myofascial pain, low back pain, peripheral neuropathy etc.
* Celiac disease or inflammatory bowel disease
* Diabetes mellitus; d) Serious mental health conditions
* Women during pregnancy or within 3 months post-partum period
* Self- reported Regular use of opioids or other illicit substances.
* Participants who have had COVID-19 should be fully recovered, and will be asked if their medical provider has made any restriction on activities.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Pain intensity and interference | Baseline and 4-week follow-up; Weekly Online Logs
  Brief Pain Inventory (BPI) scale: the 9-item scale measures pain intensity and interference using 0 - 10 rating scales. Higher score indicates higher levels of pain intensity and interference.
IBS-related symptoms | Baseline and 4-week follow-up; Weekly Online Logs
  Qualitative narrative data will be collected including self-reported stool frequency, quality, form, and abdominal bloating or distention symptoms. Online diary format data.
Electrodermal activity (EDA) | Baseline and 4-week follow-up
  EDA will be recorded non-invasively via surface electrodes on an abdominal belt; unit: µS
Electrocardiogram (ECG) | Baseline and 4-week follow-up
  ECG will be recorded non-invasively via surface electrodes on an abdominal belt; unit: mV
Electromyogram (EMG) | Baseline and 4-week follow-up
  EMG will be recorded non-invasively via surface electrodes on an abdominal belt; unit: mV
Objective integrated multimodal electrophysiological index | Baseline and 4-week follow-up
  Objective integrated multimodal electrophysiological (OIME) index as a biomarker for visceral pain will be generated and validated through integration of surface bio-signal recordings of EDA, ECG, and EMG via a supervised machine-learning algorithm.

CONTACTS AND LOCATIONS:
Locations (1):
- Vernon Cottage, Depot Campus, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No